CLINICAL TRIAL: NCT06920849
Title: Evaluation of the Influence of PRF (Platelet-rich Fibrin) on the Clinical Parameters and the Concentration of Selected Inflammation Mediators in GCF (Gingival Crevice Fluid) of Patients With Periodontitis
Acronym: PRFperio
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniBial; APK.002.122.2022 (Other: University of Bialystok)
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Periodontal Disease; Periodontitis
Keywords: periodontitis; SRP; PRF
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: The study group consisted of 20 people participants who underwent the SRP procedure (scaling and root planing) and then i-PRF was administered into the pockets. In the control group also consisting of 20 people only the SRP procedure was performed. The therapeutic procedure was performed under local anesthesia (Septanest 200, Septodont, Paris, France), using an ultrasonic device (EMS Piezon, Tip PS, EMS, Nyon, Switzerland) and hand instruments (Gracey currettes (SMS), Hu-Friedy, Chicago, IL, USA) by one operator.
  In the test group, i-PRF was prepared using a dedicated device (PRF Duo Quattro Centrifuge, Choukroun Pro-cess For PRF, Nice, France). After the SRP procedure, allocation was performed according to a randomization table prepared by a statistician, and i-PRF was administered into the pockets by one, trained operator.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRP (Experimental): In the control group (20 subjects) SRP was performed alone.
  Interventions: Procedure: SRP
- SRP+iPRF (Experimental): The test group consisted of 20 people participants who underwent the SRP procedure and then i-PRF was administered into the pockets.
  Interventions: Biological: SRP+iPRF

INTERVENTIONS:
Biological: SRP+iPRF — SRP (scaling and root planing) with iPRF (injectable platelet-rich fibrin)
  Arms: SRP+iPRF
Procedure: SRP — SRP (scaling and root planing)
  Arms: SRP

SUMMARY:
Assessment of the influence of injectable platelet-rich fibrin (i-PRF) on the clinical parameters and the inflammation mediators levels in the gingival crevicular fluid (GCF) in patients with periodontitis.

DETAILED DESCRIPTION:
Forty subjects diagnosed with periodontitis were randomly divided into two groups. In the test group, SRP was performed with the subsequent application of iPRF into periodontal pockets, while in the control group SRP was performed alone. Clinical examination was performed before and 1, 3 and 6 months after treatment. For inflammation mediators levels determination in GCF samples ELISA method will be used.

ELIGIBILITY:
Inclusion Criteria:

* clinical and radiological features of periodontitis in stage II, III or IV
* presence of at least 4 teeth and at least 2 pockets (localized not on the same tooth) with a depth of at least 5 mm in each quadrant

Exclusion Criteria:

* periodontal treatment within 3 months prior to the study;
* antibiotic therapy within 3 months prior to the study;
* smoking; presence of systemic diseases affecting periodontal healing, i.e.: immunosuppressive diseases, diabetes, osteoporosis, AIDS, hypertension treated with calcium channel blockers;
* use of steroids or other immunosuppressive drugs;
* coagulation disorders and use of drugs affecting its mechanisms;
* pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the influence of injectable platelet-rich fibrin on the clinical parameters in non-surgical treatment of periodontitis. | up to 6 months after treatment procedure
  PD (Pocket Depth) from the gingival margin to the bottom of the sulcus, measured in mm

SECONDARY OUTCOMES:
Assessment of the influence of injectable platelet-rich fibrin on the levels of inflammation mediators in the GCF in non-surgical treatment of periodontitis. | up to 3 months after treatment procedure
  Inflammation mediators level in GCF will be determined by the immunoenzymatic method ELISA (Enzyme - Linked Immunosorbent Assay) with the use of commercial kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Integrated Dentistry, Medical University of Białystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No
IPD cannot be transferred to other people due to GDPR